CLINICAL TRIAL: NCT02218840
Title: Behavioral Pharmacology Associated With Cigar Smoking
Status: Completed | Type: Observational
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 14-021CTP
Record Dates: First submitted 2014-07-30; First posted 2014-08-18 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2014-08

CONDITIONS: Cigar Smoking
Keywords: cigar smoker; smoking; behavioral pharmacology; smoking topography
MeSH Terms: conditions — Cigar Smoking; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Behavioral: Evaluation of cigar smoking topography
  Interventions: Other: Smoking topography

INTERVENTIONS:
Other: Smoking topography — Evaluation of cigar smoking topography

SUMMARY:
Lovelace Scientific Resources is conducting clinical research study for cigar smokers. This study will be evaluating the behaviors of cigar smokers and the short term effects of cigar smoking.

A cigar is defined as a cylinder of tobacco wrapped in a tobacco leaf for smoking. There are small cigars with filters that resemble cigarettes and large cigars that do not have filters. Because cigars come in so many shapes and sizes, the nicotine content varies as well. The way that a cigar smoker consumes the cigar can also have an effect on how much nicotine is absorbed. This study seeks to understand nicotine consumption and addiction in cigar smokers.

Study participation will last 1 to 4 weeks and will include 2 study-related visits. Your visits may include a physical exam, medical history review, questionnaires, blood collections, providing a urine sample, an exhaled breath test, having your vital signs collected and smoking a cigar. You will be videotaped while you smoke your cigar so that we can review the technique you use while smoking.

STUDY HYPOTHESES:

* Significant reductions in craving and withdrawal will be reported after ad libitum smoking of a cigar compared to self-report prior to cigar smoking.
* Cigar smokers will show a range of nicotine dependence, with a subset of users exceeding minimal criteria for nicotine dependence.
* Levels of nicotine, cotinine, Carbon Monoxide (CO), and 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) will increase significantly from pre- to post-cigar smoking.
* Small cigar/cigarillo users will demonstrate greater levels of dependence and greater relief from craving and withdrawal compared to large cigar users.

DETAILED DESCRIPTION:
This study seeks to better understand dependence behaviors in small and large cigar smokers. All recruited cigar smokers will be self-defined as users on ≥ 1 day(s) per week for the past 6 months. They will not be currently using any other type of tobacco product for the past 6 months. Study subjects will smoke their own type and brand of cigar upon at least 24 hours of abstinence from all tobacco products.

Dependence (both real and perceived), withdrawal relief, and craving will be measured with existing and modified behavioral scales and assessments. In addition, smoking topography (including latency to first puff, puff number, interpuff interval, and smoking duration), self-reported inhalation behaviors, and exhaled CO will also be measured.

This is a single center, un-blinded study seeking to better understand dependence behaviors in small and large cigar smokers.

Subjects will be videotaped while smoking their cigar using a digital camcorder, and the video will immediately be burned to DVD for subsequent smoking topography scoring by two separate raters. These raters will directly observe the subject during the cigar smoking exposure.

Urine samples and serial blood samples will be collected to measure biomarkers of exposure (including nicotine, cotinine, and total NNAL) before, during, and after subjects' smoking of their usual type and brand of cigar. A urine creatinine lab test will be collected pre and post exposure to correct for excreted cotinine levels. Subjects will be instructed to empty their bladders pre cigar exposure. They will then be instructed to rehydrate based on their BMI prior to the initiation of cigar smoke exposure and after 60 minutes post cigar initiation. Hepatic and renal function will be assessed at screening to determine any metabolism problems. Subjects will be asked to bring two (2) cigars of their usual type and brand. One cigar will be used to smoke; the 2nd cigar will be used to measure total nicotine content.

The cigars will be stored at ambient temperature (59º - 86º F), away from light and moisture, until analysis. Nicotine concentrations will be determined from the 2nd cigar using an analytical approach developed by Lovelace Biomedical Environmental Research Institute (LBERI). Briefly, the cigar weight will be recorded, cigar broken apart, and mixed using a mortar and pestle to create a homogenous mixture of the entire cigar. 100 mg of the cigar mixture will be weighted and nicotine extracted from the tobacco using 1mL of 50/50 dichloromethane:dichloroethane repeated twice. The extract will be evaporated and re-dissolved in 1 mL of methanol for liquid chromatography tandem mass spectrometry (LC-MS/MS) analysis.

Plasma concentrations for nicotine and cotinine will be determined using LC-MS/MS and values exported to Phoenix WinNonlin for pharmacokinetic analysis. Plasma Tmax and Cmax will be reported using a table in a word document and in figures generated using WinNonlin. The amount of cotinine and total NNAL excreted will be reported by determining the urinary concentration of each compound by LC-MS/MS analysis and multiplying the determined concentration by the total volume of urine recovered. Individual data along with grouped results will be reported. The pharmacokinetic data will be provided to the sponsor after uploading to SAS.

The subjects will be cigar smokers who are not seeking treatment for smoking cessation and who are not currently using any other type of tobacco, but may be former users. They must agree to abstain from smoking for at least 24 hours prior to the exposure day and will be informed that they must remain abstinent from all forms of tobacco including nicotine patches, gum, etc. Abstinence will be verified at the beginning of the test day through expired CO and self-report. While it could be desirable to use urinary cotinine levels as a further marker of abstinence, urinary cotinine levels do not appear to reach undetectable levels in smokers after 24 hours. Instead, in regular smokers, negligent levels are reached only after abstinence of 7-8 days, which would place significant burden on subjects for this study. All subjects should be healthy males and females, 18 years of age or older, with no self-reported psychiatric illnesses that would interfere with the subjects ability to complete the session (i.e. schizophrenia, severe depression).

Women who are pregnant (as verified by a urine pregnancy test at Visit 1 and 2) or breastfeeding will be excluded.

Subjects will be asked questions concerning the type and quantity of prescribed and non-prescribed drugs that they are currently using. If, as a result of the screening, the subject is determined to be ineligible to continue participation in the study, he/she will be excused from further participation. A target of sixty four (64) completed subjects will be recruited to ensure sufficient statistical power to test main effects across the following groups:

1. Primary vs. secondary cigar users
2. Self-reported inhaling behavior vs. self-reported non-inhaling behavior
3. Small cigar (including cigarillos) vs. large cigar (including premium) users
4. White vs. non-white adults
5. Male vs. Female adults A power analysis was conducted to determine the overall sample size needed to test the main effects above. According to this power analysis (see below), the study will require 64 subjects assuming a balanced design across each of the above factors (i.e. subjects are stratified across the 5 factors for a total of 32 groups). However, given the potential difficulty in filling each group of the above design, we may recruit up to 50% more subjects (i.e. 96), which will ensure that each of the above groups are sufficiently represented in the final sample. Finally, assuming a 10% dropout rate, an additional 10 subjects may be enrolled for a total sample size of 106.

Subjects will be monitored for adverse events (AEs) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Willing to voluntarily sign the IRB approved informed consent form (ICF)
* Willing to complete all the requirements of the study
* Male or Female, ≥ 18 years of age
* Female subjects must be either:

Surgically sterile defined as having had a hysterectomy, bilateral oophorectomy, or tubal ligation, amenorrheic for at least two years prior to screening visit, or otherwise incapable of becoming pregnant Or Willing to practice an effective method of birth control if sexually active, taking hormonal prescription oral contraceptives, progesterone implants or injections, contraceptive patch, intrauterine device, or male partner with a vasectomy. A double barrier method such as condoms, diaphragms, or cervical caps with spermicidal foam, cream, or gel, or abstinence may be used as a method of birth control

* Must be either a primary cigar or a secondary cigar smoker. Must have a self-reported history of using cigars on ≥1 day per week for the past 6 months
* Primary cigar users must report no significant prior use of cigarettes (< 100 cigarettes in lifetime and no use of cigarettes in the past 6 months)
* Secondary cigar users must self-report regular use of cigarettes in the past before making the switch to cigars, and must report no use of cigarettes in the past 6 months
* Must be able to self-report inhaling behavior as either inhaler or non-inhaler
* Must be able to identify primary type of cigars smoked as either small cigar (including cigarillos), large cigars, or premium cigars
* English-speaking volunteers who are not seeking treatment for smoking cessation at the time of the study
* Have an exhaled carbon monoxide (CO) level of <10 ppm at visit 2
* Demonstrate no clinically significant contraindications for study participation, in the judgment of the Principal Investigator

Exclusion Criteria:

* Women of Child Bearing Potential (WOCBP) with a positive urine human chorionic gonadotropin (Urine β- hCG) pregnancy test within 10 days prior to Visit 2
* Pregnant and/or nursing females
* Use of any other type tobacco product (except cigars), non-tobacco nicotine-containing product(s), smoking cessation medications, such as varenicline (Chantix®) and bupropion (Zyban®), or NRT (Nicotine Replacement Therapy) within 60 days of study enrollment
* Have any previous self-reported medical adverse reaction to nicotine or tobacco, (for example nausea, headache and chest pain)
* Subjects who self-report a clinically significant concomitant disease or illness at either screening or visit 2, including but not limited to depression, schizophrenia, uncontrolled respiratory or cardiovascular disease, which in the opinion of the Principal Investigator or designee would preclude safe and /or successful completion of this study
* Subject demonstrates an elevated liver function of ≥ 2 times the upper limit of normal at screening
* Subject demonstrates an elevated renal function of ≥ 2 times the upper limit of normal at screening
* Subject intends to stop smoking cigars in the next month
* Unwilling to abstain from cigar smoking and all tobacco and nicotine use for at least 24 hours prior to exposure, Visit 2

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be cigar smokers who are not seeking treatment for smoking cessation and who are not currently using any other type of tobacco, but may be former users.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-01-08 (Actual); Study Completion 2016-03-02 (Actual)

PRIMARY OUTCOMES:
Assess Beharioral/Self-Reported Aspects of Cigar Smoking | 4 weeks
  Characterize and quantify dependence, withdrawal relief, cravings, puff topography

SECONDARY OUTCOMES:
Evaluate smoking exposure | 4 weeks
  Identifying smoking puff topography and laboratory markers of exposure (nicotine, NNAL, breath CO, and cotinine).

CONTACTS AND LOCATIONS:
Overall Officials: Michael R McGuire, MD, Principal Investigator — Lovelace Scientific Resources, Inc
Locations (1):
- Lovelace Scientific Resources, Inc, Albuquerque, New Mexico, United States